CLINICAL TRIAL: NCT02646137
Title: Comparison of Single Session Transarterial Chemoembolization Combined With Microwave Ablation or Radiofrequency Ablation in Treatment of Hepatocellular Carcinoma: A Randomized Controlled Study
Brief Title: Single Session Combined Locoregional Therapies for Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Consultant liver and GIT diseases- Tanta university hospital, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Combined TACE and RF
Record Dates: First submitted 2016-01-01; First posted 2016-01-05 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Transarterial chemoembolization (TACE) (Active Comparator): treated by transarterial chemoembolization
  Interventions: Drug: Transarterial chemoembolization (TACE)
- Radiofrequency ablation with TACE (Experimental): Radiofrequency ablation combined with TACE
  Interventions: Procedure: Radiofrequency ablation combined with TACE
- Microwave ablation combined with TACE (Experimental): Microwave ablation combined with TACE.
  Interventions: Procedure: Microwave ablation combined with TACE

INTERVENTIONS:
Drug: Transarterial chemoembolization (TACE) — TACE exploits the preferential hepatic arterial supply of liver tumors for targeted delivery of chemotherapeutic agents followed by embolization or reduction in arterial flow using various types of particles
  Other Names: Transarterial chemoembolization
  Arms: Transarterial chemoembolization (TACE)
Procedure: Radiofrequency ablation combined with TACE — Radiofrequency ablation (RFA) is an alternative therapy for HCC and liver metastases that can destroy a tumor by inducing thermal injury to the tissue through electromagnetic energy deposition
  Arms: Radiofrequency ablation with TACE
Procedure: Microwave ablation combined with TACE — Microwave ablation (MWA) is an appealing alternative therapy for HCC in which a microwave antenna is placed directly into the tumor, emitting an electromagnetic wave which agitates water molecules in the surrounding tissue, producing friction and heat, thereby inducing cell death via coagulation necrosis
  Arms: Microwave ablation combined with TACE

SUMMARY:
Hepatocellular carcinoma is the third most common cause of cancer-related mortality. In recent years, transarterial chemoembolization, radio frequency ablation and microwave ablation have been accepted as treatment modalities for patients with surgically unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
To compare between combination treatment with radiofrequency or microwave ablation followed by transarterial chemoembolization and performed in a single session.

ELIGIBILITY:
Inclusion Criteria:

* Child classification A or B.
* serum albumin ≥ 3 gm/L.
* serum bilirubin < 2.5 mg/dL.
* platelet count ≥70,000 mm3.
* INR ≤ 1.6.
* serum creatinine < 2 mg/dl.
* tumor size more than 4 cm and confined to one lobe of the liver.

Exclusion Criteria:

* Patients with portal vein thrombosis.
* A technically inaccessible hepatic artery.
* Metastatic HCC.
* More than three lesions.
* lesions in close proximity to the portal vein (PV),inferior vena cava (IVC) or gall bladder were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful ablation | 3 months
  The total number of patients with successful ablation

CONTACTS AND LOCATIONS:
Overall Officials: Elshazly Sheta, Professor, Principal Investigator — Hepatology and gastroenterology dept.-Tanta; Ferial El-kalla, Professor, Principal Investigator — Division of Gastroenterology and Hepatology- Tanta; Mohamed Elgharib, Professor, Study Director — Interventional radiology - Ainshams university- Egypt; Abdelrahman kobtan, Consultant, Study Chair — liver diseases dept.-Tanta university hospital; Mohamed Elhendawy, Consultant, Study Chair — liver diseases dept.-Tanta university hospital; Sherief Abd-Elsalam, Consultant, Study Chair — Hepatology and gastroenterology dept.-Tanta; Ibrahim Amer, Consultant, Study Chair — Liver diseases and gastroenterology dept.-Tanta university hospital
Locations (1):
- Tanta university hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided